CLINICAL TRIAL: NCT04884737
Title: Decreasing Intraoperative Skin Damage in Prone Position Surgeries
Acronym: P3I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Barbara Bates-Jensen, PhD, RN, FAAN, Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 21-000240
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Pressure Injury
MeSH Terms: conditions — Pressure Ulcer | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: In months 1-3 Pre-Intervention participants will have 6 skin assessments at face (chin, cheeks, forehead), chest, and iliac crest: preoperative, Post Anesthesia Recovery Unit, transfer to floor, and post-operative days 1, 3 and 5.
  In months 4-6 Intervention participants will have the same skin assessments at the same times and will have the dressings placed pre-operatively and removed following surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pre-Intervention (No Intervention): Pre-Intervention Group participants will have 6 visits. During the pre-intervention baseline (3 months) participants will undergo visual skin assessment and SEM Scanner readings at face (chin, cheeks, forehead), chest, and iliac crest, conducted by the research staff: 1.) consent and preoperative, 2.) immediately following surgery in the Post Anesthesia Recovery (PAR) Unit, 3.) on transfer to the floor unit, 4.) post-operative day 1, 5.) post-operative day 3 and 6.) post-operative day 5 or discharge from hospital (whichever occurs first). Combined visit time will be 1 hour and 40 minutes.
- Intervention (Experimental): Intervention Group participants will have 7 visits. During intervention (3 months) research staff will conduct the visual skin assessment and SEM Scanner readings at face (chin, cheeks, forehead), chest, and iliac crest, and place the MBF dressings to the face (chin, cheeks, forehead), chest and iliac crest: 1.consent and preoperative, 2. MBF dressing placement, 3.) immediately following surgery in the PAR unit with the MBF dressings removed , 4.) on transfer to the floor unit, 5.) post-operative day 1, 6.) post operative day 3 and 7.) post-operative day 5 or discharge from hospital (whichever occurs first). Combined visit time will be 1 hour and 55 minutes.
  Interventions: Other: Mepilex Border Flex® (MBF) dressing

INTERVENTIONS:
Other: Mepilex Border Flex® (MBF) dressing — A new dressing technology (Mepilex Border Flex® (MBF)) provides increased conformability of the dressing to the skin with the ability of the dressing to move in all directions (e.g., 360-degree flexibility) with even slight body movements. Limited data exists on use of silicone foam dressings with all direction flexibility during prone surgical procedures.
  Arms: Intervention

SUMMARY:
Preventing Pressure Injuries among patients undergoing spinal or orthopedic surgery in the prone position is challenging because of position required for surgical access and limited availability of pressure reduction surfaces for prone position operating tables. A new dressing technology (Mepilex Border Flex® (MBF) provides increased conformability of the dressing to the skin with the ability of the dressing to move in all directions (e.g., 360-degree flexibility) with even slight body movements. Limited data exists on use of silicone foam dressings with all direction flexibility during prone surgical procedures.

The investigators will partents scheduled for surgery in the prone position at UCLA Santa Monica Medical Center and propose to examine use of the MBF dressings on the chest, iliac crest, and face (chin, cheeks, forehead) of patients undergoing this type of surgery using a prospective, non-randomized pre/post intervention clinical trial design.

Three outcome measures will be compared between patients undergoing prone surgery with standard care (no dressings, pressure reduction positioning on the operating table) and those with standard care and use of MBF dressings placed on the chest, iliac crest and face: (1) incidence of erythema and pressure injuries on face, chest and iliac crest determined by visual skin assessment between the two groups, (2) incidence of moisture associated skin damage (MASD) and friction abrasions on face, chest and iliac crest determined by visual skin assessment between the two groups, and (3) SEM measures indicative of pressure injury damage on face, chest, iliac crest between the two groups.

The study will also include a 6-month retrospective medical record review of patients who underwent prone surgeries from February 1, 2018 through July 31, 2018 to determine a historical pressure injury facility incident rate. The year 2018 was chosen to avoid changes associated with the COVID-19 pandemic.

DETAILED DESCRIPTION:
Preventing pressure injuries (PrIs) from developing during surgery is difficult due to insensitivity and immobility of the patient and the positioning needed for safe surgical access. Intraoperative acquired pressure injury (IAPI) rates are reported from 4% to 45% (1). IAPI rates vary due to differences in defining PrIs, surgical positions and because tissue damage that occurs in surgery may not be visible on the skin surface initially with the resulting PrI presenting several days post operatively (2,3). The sustained pressure, deformation, and shear forces on the tissues combined with changes in blood flow due to blood loss, vasopressor and anesthesia use, and temperature changes present unique risk factors for PrI development during surgery (1). Reducing PrI damage during surgery requires preventive strategies to decrease the mechanical forces of pressure and shear on the tissues loaded in the unique positions required for surgical access. In the supine position for surgery, use of silicone foam dressings on the sacrum and heels with pressure reducing devices on the operating table have decreased IAPIs (4, 5).

The prone position for surgery has been shown to be a risk factor for IAPIs in multiple studies (1,2,4,14). Yet, there is limited data on IAPIs for surgeries in the prone position with Luo and colleagues reporting incidence at 4.7% and Yoshimura et al showing an 11% incidence (4,15). Preventing PrIs among patients undergoing spinal or orthopedic surgery in the prone position is especially challenging because of positioning required for surgical access and limited availability of pressure reduction surfaces for prone positioner operating tables (2,15). The face, chest, and iliac crest are all loaded on small operating table surfaces in the prone position. These anatomic locations have limited soft tissue for compression and small surface areas and because of this, distribution of pressure and shear forces over a large surface area is not possible. Thus, the intensity of the pressure and shear force over these anatomic areas is high. Shear force is particularly problematic as tissues change due to variations in blood volume and flow, anesthesia and vasopressor use, and initiation of the inflammatory response during the surgical procedure all of which may increase shear forces on the tissues (1,2,16). Use of silicone foam dressings on the iliac crest and chest has been shown to reduce IAPIs in the prone position for spinal surgery (15). Most recently, use of silicone foam dressings has been suggested for use to decrease PrIs in patients with acute respiratory distress syndrome (ARDS) from COVID-19 who are placed in prone position to manage respiratory distress (17,18). Issues with use of silicone foam dressings intraoperatively is keeping the dressing in place while positioning for surgery preoperatively, protecting the skin and allowing for movement and changes in the tissues intraoperatively, and safe nontraumatic removal immediately postoperatively. A new dressing technology (Mepilex Border Flex® (MBF)) provides increased conformability of the dressing to the skin with the ability of the dressing to move in all directions (e.g., 360-degree flexibility) with even slight body movements while using a silicone-based adhesive allowing for atraumatic removal.

The investigators will examine use of MBF dressings on the chest, iliac crest, and face (chin, cheeks, forehead) of patients undergoing surgery in a prone position using a prospective, non-randomized pre/post-intervention clinical trial. The specific aims are to:

1. Compare IAPI, erythema, and skin damage (e.g., friction abrasions, moisture associated skin damage (MASD)) incidence of patients undergoing surgery in a prone position with use of standard care to use of MBF dressings placed on chest, iliac crest, and face with standard care.
2. Compare subepidermal moisture (SEM) values (a biophysical measure of inflammatory tissue changes) of patients undergoing surgery in a prone position with use of standard care to use of MBF dressings placed on chest, iliac crest, and face along with standard care.
3. Explore cost estimates for use of MBF dressings placed on chest, iliac crest, and face for surgery in a prone position.

Three outcome measures will be compared between patients undergoing prone surgery with standard care (no dressings, pressure reduction positioning on the operating table) and those with standard care and use of MBF dressings placed on chest, iliac crest, and face: (1) incidence of erythema and PrIs on anatomic locations from visual skin assessment, (2) incidence of moisture associated skin damage (MASD) and friction abrasions on anatomic locations, and (3) SEM measures indicative of PrI damage.

The investigators will also complete a 6-month retrospective medical record review of patients who underwent prone surgeries from February 1, 2018 through July 31, 2018 to determine a historical PrI facility incidence rate. The year 2018 was chosen to avoid changes associated with the COVID-19 pandemic.

The investigators will obtain written informed consent to participate in the study directly from patients who are able to provide informed consent.

Participants will be recruited from patients in the neurological and the orthopedic surgery groups scheduled for prone surgery UCLA Santa Monica Medical Center. Participant inclusion criteria are over 18 years of age and able to provide informed self-consent. Exclusions to participation include less than 18 years old, inability to provide informed consent, and scheduled for surgery in a position other than prone position.

The study data collection period is anticipated to be 6 months, 3 months of pre-intervention baseline assessments followed by 3 months of intervention assessments.

During pre-intervention baseline (3 months) participants will undergo visual skin assessment and SEM Scanner readings at face (chin, cheeks, forehead), chest and iliac crest, conducted by the research staff, preoperatively, immediately following surgery in the Post Anesthesia Recovery (PAR) Unit, on transfer to the floor unit, post-operative day 3 and post-operative day 5 or discharge from hospital (whichever occurs first).

During intervention (3 months) participants will undergo visual skin assessment and SEM Scanner readings at face (chin, cheeks, forehead), chest and iliac crest, and then placement of MBF dressings to the face, chest and iliac. MBF dressings will be removed in the PAR unit, on transfer to the floor unit, post-operative day 3 and post-operative day 5 or discharge from hospital (whichever occurs first).

Research staff will collect all data after training in all protocols by the PI. Data collection includes medical record abstraction, visual skin assessments, and SEM Scanner measures. Each is described below.

The electronic medical record will be abstracted for demographic data (gender, age, race/ethnicity) and medical data (height, weight, body mass index, comorbidities such as diabetes, hypertension, peripheral vascular disease and, smoking status, medical diagnoses, Braden Scale for predicting Pressure Sores (Braden) score, use of any PrI preventive strategies such as support surface use, repositioning schedules), surgery type, surgery length, use of vibration machines or other instruments in surgery, length of time in PAR unit, anesthesia used, use of vasopressors during surgery, estimated blood loss, volume of fluids provided during surgery, blood pressure during surgery, American Society of Anesthesiologists physical status score and documentation of any skin damage including PrIs, MASD, and friction abrasions.

A 6-month retrospective medical record review of patients who underwent prone surgery between February 1, 2018 through July 31, 2018 will be done to determine the historical PrI incidence for UCLA Santa Monica Medical Center. The retrospective medical record review will include data as noted above.

Visual skin assessment training of research staff will emphasize stage 1 PrIs and deep tissue injury (DTI) Research staff will assess skin health through direct visual assessments preoperatively or within 1 week of scheduled surgery, immediately after surgery in PAR unit, on transfer to the floor unit, post-operative days 3 and 5 or discharge whichever occurs first. Participants will be positioned in bed in a supine position for visual assessments. Eight anatomic locations will be assessed: right and left chest at nipple line, iliac crest, and cheeks, mid forehead and chin. Skin will be assessed for discoloration (redness), erythema, PrI, MASD, and friction abrasion. Areas of visual skin discoloration will be palpated for blanchability using finger palpation and defined as blanchable versus non-blanchable. Erythema will be graded as minimal, moderate, or severe discoloration. DTI will be defined as severe skin discoloration (purple or maroon in light skin tones and black to blue-grey in dark skin tones) with or without blanching. Stage 1 PrIs will be defined as moderate skin discoloration (all skin tones), with non-blanching (non dark skin tones). PrIs more severe than stage 1 will be classified using the EPUAP/NPIAP/PPPIA's 2019 staging system (1) and assessed using the Bates-Jensen Wound Assessment Tool (BWAT) (32).

The SEM readings will be obtained on clean dry skin directly over each anatomic location using the SEM Scanner (Bruin Biometrics, Los Angeles, CA), a handheld dermal phase meter that requires light skin touch and provides SEM readings in 3 seconds (range 0-7 picoFarads (pF)) concurrently with the visual skin assessments. The SEM Scanner uses dielectric parameters, high-frequency low power electromagnetic waves of 32 kHz are transmitted via an electrode that is manually placed on the skin surface. In the skin, the induced electrical field interacts mainly with water molecules closest to the electrode with depth of interaction depending on the diameter of the circular electrode (in this study at a depth of 4mm) (19-21). The portion of the electromagnetic energy that is not absorbed by tissue water is reflected and measured by the device and displayed in the measuring unit. SEM values are displayed in picoFarads. Reliability of the device has been previously reported (33).

Descriptive statistics will be used to describe the sample. Chi square (categorical data), t-tests (continuous data) and Analysis of Variance (ANOVA) will be used as appropriate to compare demographic and medical data between the two study groups and to compare the total sample to the retrospective historical sample.

Costs of the dressings will be described.

ELIGIBILITY:
Inclusion Criteria:

* A participant must 18 years or older and is scheduled for surgery in the prone position to be conducted at UCLA Santa Monica Medical Center.

Exclusion Criteria:

* Patients who are not scheduled for surgery in the prone position. Patients with known allergy to the components of the Mepilex Border Flex (MBF) dressing which consists of silicone, polyurethane, polyacrylate, viscose, polyester and polyolefin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Santa Monica Medical Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. European Pressure Ulcer Advisory Panel, National Pressure Injury Advisory Panel and Pan Pacific Pressure Injury Alliance. Prevention and Treatment of Pressure Ulcers/Injuries: Clinical Practice Guideline. The International Guideline. Emily Haesler (Ed.). EPUAP/NPIAP/PPPIA: 2019.
- [Background] Gefen A, Creehan S, Black J. Critical biomechanical and clinical insights concerning tissue protection when positioning patients in the operating room: A scoping review. Int Wound J. 2020 Oct;17(5):1405-1423. doi: 10.1111/iwj.13408. Epub 2020 Jun 4. PMID 32496025
- [Background] Spector WD, Limcangco R, Owens PL, Steiner CA. Marginal Hospital Cost of Surgery-related Hospital-acquired Pressure Ulcers. Med Care. 2016 Sep;54(9):845-51. doi: 10.1097/MLR.0000000000000558. PMID 27219637
- [Background] Luo M, Long XH, Wu JL, Huang SZ, Zeng Y. Incidence and Risk Factors of Pressure Injuries in Surgical Spinal Patients: A Retrospective Study. J Wound Ostomy Continence Nurs. 2019 Sep/Oct;46(5):397-400. doi: 10.1097/WON.0000000000000570. PMID 31513127
- [Background] Bulfone G, Bressan V, Morandini A, Stevanin S. Perioperative Pressure Injuries: A Systematic Literature Review. Adv Skin Wound Care. 2018 Dec;31(12):556-564. doi: 10.1097/01.ASW.0000544613.10878.ed. PMID 30475284
- [Background] Bulfone G, Marzoli I, Quattrin R, Fabbro C, Palese A. A longitudinal study of the incidence of pressure sores and the associated risks and strategies adopted in Italian operating theatres. J Perioper Pract. 2012 Feb;22(2):50-6. doi: 10.1177/175045891202200202. PMID 22724304
- [Background] Schoonhoven L, Defloor T, Grypdonck MH. Incidence of pressure ulcers due to surgery. J Clin Nurs. 2002 Jul;11(4):479-87. doi: 10.1046/j.1365-2702.2002.00621.x. PMID 12100644
- [Background] Hayes RM, Spear ME, Lee SI, Krauser Lupear BE, Benoit RA, Valerio R, Dmochowski RR. Relationship between time in the operating room and incident pressure ulcers: a matched case-control study. Am J Med Qual. 2015 Nov-Dec;30(6):591-7. doi: 10.1177/1062860614545125. Epub 2014 Jul 30. PMID 25077711
- [Background] Yoshimura M, Iizaka S, Kohno M, Nagata O, Yamasaki T, Mae T, Haruyama N, Sanada H. Risk factors associated with intraoperatively acquired pressure ulcers in the park-bench position: a retrospective study. Int Wound J. 2016 Dec;13(6):1206-1213. doi: 10.1111/iwj.12445. Epub 2015 Jun 4. PMID 26043765
- [Background] Riemenschneider KJ. Prevention of Pressure Injuries in the Operating Room: A Quality Improvement Project. J Wound Ostomy Continence Nurs. 2018 Mar/Apr;45(2):141-145. doi: 10.1097/WON.0000000000000410. PMID 29521925
- [Background] de Oliveira KF, Nascimento KG, Nicolussi AC, Chavaglia SRR, de Araujo CA, Barbosa MH. Support surfaces in the prevention of pressure ulcers in surgical patients: An integrative review. Int J Nurs Pract. 2017 Aug;23(4). doi: 10.1111/ijn.12553. Epub 2017 Jun 23. PMID 28643855
- [Background] Joseph J, McLaughlin D, Darian V, Hayes L, Siddiqui A. Alternating Pressure Overlay for Prevention of Intraoperative Pressure Injury. J Wound Ostomy Continence Nurs. 2019 Jan/Feb;46(1):13-17. doi: 10.1097/WON.0000000000000497. PMID 30601427
- [Background] Strauss R, Preston A, Zalman DC, Rao AD. Silicone Foam Dressing for Prevention of Sacral Deep Tissue Injuries Among Cardiac Surgery Patients. Adv Skin Wound Care. 2019 Mar;32(3):139-142. doi: 10.1097/01.ASW.0000553111.55505.84. PMID 30801352
- [Background] Gao L, Yang L, Li X, Chen J, Du J, Bai X, Yang X. The use of a logistic regression model to develop a risk assessment of intraoperatively acquired pressure ulcer. J Clin Nurs. 2018 Aug;27(15-16):2984-2992. doi: 10.1111/jocn.14491. Epub 2018 Jun 5. PMID 29679411
- [Background] Yoshimura M, Ohura N, Tanaka J, Ichimura S, Kasuya Y, Hotta O, Kagaya Y, Sekiyama T, Tannba M, Suzuki N. Soft silicone foam dressing is more effective than polyurethane film dressing for preventing intraoperatively acquired pressure ulcers in spinal surgery patients: the Border Operating room Spinal Surgery (BOSS) trial in Japan. Int Wound J. 2018 Apr;15(2):188-197. doi: 10.1111/iwj.12696. Epub 2016 Dec 7. PMID 27928911
- [Background] Dharmavaram S, Jellish WS, Nockels RP, Shea J, Mehmood R, Ghanayem A, Kleinman B, Jacobs W. Effect of prone positioning systems on hemodynamic and cardiac function during lumbar spine surgery: an echocardiographic study. Spine (Phila Pa 1976). 2006 May 20;31(12):1388-93; discussion 1394. doi: 10.1097/01.brs.0000218485.96713.44. PMID 16721305
- [Background] Peko L, Barakat-Johnson M, Gefen A. Protecting prone positioned patients from facial pressure ulcers using prophylactic dressings: A timely biomechanical analysis in the context of the COVID-19 pandemic. Int Wound J. 2020 Dec;17(6):1595-1606. doi: 10.1111/iwj.13435. Epub 2020 Jul 3. PMID 32618418
- [Background] Moore Z, Patton D, Avsar P, McEvoy NL, Curley G, Budri A, Nugent L, Walsh S, O'Connor T. Prevention of pressure ulcers among individuals cared for in the prone position: lessons for the COVID-19 emergency. J Wound Care. 2020 Jun 2;29(6):312-320. doi: 10.12968/jowc.2020.29.6.312. PMID 32530776
- [Background] Nuutinen J, Ikaheimo R, Lahtinen T. Validation of a new dielectric device to assess changes of tissue water in skin and subcutaneous fat. Physiol Meas. 2004 Apr;25(2):447-54. doi: 10.1088/0967-3334/25/2/004. PMID 15132310
- [Background] Alanen E, Nuutinen J, Nicklen K, Lahtinen T, Monkkonen J. Measurement of hydration in the stratum corneum with the MoistureMeter and comparison with the Corneometer. Skin Res Technol. 2004 Feb;10(1):32-7. doi: 10.1111/j.1600-0846.2004.00050.x. PMID 14731246
- [Background] Palenske J, Morhenn VB. Changes in the skin's capacitance after damage to the stratum corneum in humans. J Cutan Med Surg. 1999 Jan;3(3):127-31. doi: 10.1177/120347549900300304. PMID 10082592
- [Background] Bates-Jensen BM, McCreath HE, Pongquan V, Apeles NC. Subepidermal moisture differentiates erythema and stage I pressure ulcers in nursing home residents. Wound Repair Regen. 2008 Mar-Apr;16(2):189-97. doi: 10.1111/j.1524-475X.2008.00359.x. PMID 18318804
- [Background] Bates-Jensen BM, McCreath HE, Kono A, Apeles NC, Alessi C. Subepidermal moisture predicts erythema and stage 1 pressure ulcers in nursing home residents: a pilot study. J Am Geriatr Soc. 2007 Aug;55(8):1199-205. doi: 10.1111/j.1532-5415.2007.01261.x. PMID 17661958
- [Background] Bates-Jensen BM, McCreath HE, Pongquan V. Subepidermal moisture is associated with early pressure ulcer damage in nursing home residents with dark skin tones: pilot findings. J Wound Ostomy Continence Nurs. 2009 May-Jun;36(3):277-84. doi: 10.1097/WON.0b013e3181a19e53. PMID 19448508
- [Background] Guihan M, Bates-Jenson BM, Chun S, Parachuri R, Chin AS, McCreath H. Assessing the feasibility of subepidermal moisture to predict erythema and stage 1 pressure ulcers in persons with spinal cord injury: a pilot study. J Spinal Cord Med. 2012 Jan;35(1):46-52. doi: 10.1179/204577211X13209212104141. PMID 22330190
- [Background] Bates-Jensen BM, McCreath HE, Patlan A. Subepidermal moisture detection of pressure induced tissue damage on the trunk: The pressure ulcer detection study outcomes. Wound Repair Regen. 2017 May;25(3):502-511. doi: 10.1111/wrr.12548. Epub 2017 May 31. PMID 28494507
- [Background] Bates-Jensen BM, McCreath HE, Nakagami G, Patlan A. Subepidermal moisture detection of heel pressure injury: The pressure ulcer detection study outcomes. Int Wound J. 2018 Apr;15(2):297-309. doi: 10.1111/iwj.12869. Epub 2017 Dec 17. PMID 29250926
- [Background] Gefen A, Gershon S. An Observational, Prospective Cohort Pilot Study to Compare the Use of Subepidermal Moisture Measurements Versus Ultrasound and Visual Skin Assessments for Early Detection of Pressure Injury. Ostomy Wound Manage. 2018 Sep;64(9):12-27. PMID 30256748
- [Background] Smith G. Improved clinical outcomes in pressure ulcer prevention using the SEM scanner. J Wound Care. 2019 May 2;28(5):278-282. doi: 10.12968/jowc.2019.28.5.278. PMID 31067157
- [Background] Okonkwo H, Bryant R, Milne J, Molyneaux D, Sanders J, Cunningham G, Brangman S, Eardley W, Chan GK, Mayer B, Waldo M, Ju B. A blinded clinical study using a subepidermal moisture biocapacitance measurement device for early detection of pressure injuries. Wound Repair Regen. 2020 May;28(3):364-374. doi: 10.1111/wrr.12790. Epub 2020 Jan 21. PMID 31965682
- [Background] O'Brien G, Moore Z, Patton D, O'Connor T. The relationship between nurses assessment of early pressure ulcer damage and sub epidermal moisture measurement: A prospective explorative study. J Tissue Viability. 2018 Nov;27(4):232-237. doi: 10.1016/j.jtv.2018.06.004. Epub 2018 Jun 25. PMID 30017215
- [Background] Bates-Jensen BM, McCreath HE, Harputlu D, Patlan A. Reliability of the Bates-Jensen wound assessment tool for pressure injury assessment: The pressure ulcer detection study. Wound Repair Regen. 2019 Jul;27(4):386-395. doi: 10.1111/wrr.12714. Epub 2019 Mar 18. PMID 30828890
- [Background] Clendenin M, Jaradeh K, Shamirian A, Rhodes SL. Inter-operator and inter-device agreement and reliability of the SEM Scanner. J Tissue Viability. 2015 Feb;24(1):17-23. doi: 10.1016/j.jtv.2015.01.003. Epub 2015 Feb 3. PMID 25682271
- [Derived] Bates-Jensen BM, Crocker J, Nguyen V, Robertson L, Nourmand D, Chirila E, Laayouni M, Offendel O, Peng K, Romero SA, Fulgentes G, McCreath HE. Decreasing Intraoperative Skin Damage in Prone-Position Surgeries. Adv Skin Wound Care. 2024 Aug 1;37(8):413-421. doi: 10.1097/ASW.0000000000000186. PMID 39037095

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-Intervention | Intervention
Started | 50 | 57
Completed | 39 | 48
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Intervention | Intervention | Total
Number analyzed (Participants) | 39 | 48 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (14.4) | 59.5 (16.3) | 61.0 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 22 | 31 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 37 | 41 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 28 | 34 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 48 | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intraoperative Acquired Pressure Injuries (IAPI)
Description: Pressure damage to skin and soft tissues based on visual skin assessment
Time Frame: Within 5 days of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention | Intervention
Number analyzed (Participants) | 39 | 48
Participants | 13 | 14

2. Primary Outcome: Number of Participant With Erythema, Abrasions, and Moisture Associated Skin Damage (MASD)
Description: redness and skin damage from moisture or friction
Time Frame: Within 5 days of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention | Intervention
Number analyzed (Participants) | 39 | 48
Participants | 0 | 0

3. Primary Outcome: Number of Participants With a (Sub-epidermal Moisture) SEM Scanner Difference of Greater Than 0.5pF Measured at Preoperative Day of Surgery and at Least One Postoperative Assessment
Description: Difference of greater than 0.5pF between pre-operative and first post-operative readings of SEM (sub epidermal moisture or edema) at any anatomic site (face sites, chest, iliac crest)
Time Frame: preoperatively and first postoperative assessment (within 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention | Intervention
Number analyzed (Participants) | 39 | 48
Participants | 17 | 11

ADVERSE EVENTS:
Time Frame: up to 5 days post surgery
Arm/Group | Pre-Intervention | Intervention
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/48
Other Adverse Events (participants affected / at risk) | 0/39 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04884737/Prot_SAP_000.pdf